CLINICAL TRIAL: NCT02023190
Title: Changes in Body Composition and Nutritional Status Assessed by Bioelectrical Impedance Vector Analysis in Cirrhotic Patients Undergoing Liver Transplantation
Brief Title: Changes in Body Composition and Nutritional Status in Patients Undergoing Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: LT01
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; liver transplant; nutritional status; bioelectrical impedance vector analysis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nutritional assessment: Nutritional assessment will be performed by bioelectrical impedance vector analysis

SUMMARY:
Liver transplant is the goal treatment for every patient with end-stage chronic liver disease.

Quality of life improves after transplant because the main complications of end-stage liver disease disappear, but due to immunosuppression other alterations appear such as metabolic alterations, weight gain, among others.

Body composition and nutritional status can be affected do to post-transplant pharmacologic therapy.

DETAILED DESCRIPTION:
Body composition and nutritional status can be affected due to post-transplant pharmacologic therapy.

This is a prospective cohort study, patients from liver transplant waiting list will be assessed, pre and post-transplant measures of body composition and nutritional status will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis (any etiology)
* Enrolled in waiting list for tliver transplant

Exclusion Criteria:

* Hepatocellular carcinoma
* Chronic renal failure
* Congestive cardiac failure
* Extremity amputation
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be selected from the transplant enrollment list at the Department of Gastroenterology in a tertiary care center in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Body composition | Baseline, 7 days, 1 month, 3 months and 6 months post-tranpslant
  Body composition will be assessed through bioelectrical impedance vector analysis graph.

SECONDARY OUTCOMES:
Liver function tests | Baseline, 7 days, 1 month, 3 months and 6 months post-tranpslant

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD MSci, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Astrid Ruiz-Margáin, M.Sci, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico